CLINICAL TRIAL: NCT00310492
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Parallel Group Study to Demonstrate the Efficacy of a 12-month Subcutaneous Specific Immunotherapy With ALK-depot SQ Milbenmischung in Patients With Atopic Dermatitis and Proven IgE-mediated Sensitization to House Dust Mites
Brief Title: Efficacy and Safety Trial of ALK-depot SQ Mites in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHX0556
Record Dates: First submitted 2006-04-02; First posted 2006-04-04 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous immunotherapy (Active Comparator): Subcutaneous injections with ALK-depot SQ mites to 100,000 SQ-U
  Interventions: Biological: subcutaneous immunotherapy
- Subcutaneous injections (Placebo Comparator): placebo injections
  Interventions: Biological: subcutaneous immunotherapy

INTERVENTIONS:
Biological: subcutaneous immunotherapy — Updosing by 16 injections to 100,000 SQ-U
  Other Names: ALK-depot SQ mites

SUMMARY:
This trial is performed to assess the efficacy and safety of ALK-depot SQ mites for treatment of atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Positive specific IgE to house dust mites
* Atopic dermatitis according to Hanifin/Rajka
* Chronic course of Atopic dermatitis
* SCORAD larger than 25 points

Exclusion Criteria:

* Erythrodermia
* Syst.treatment with gcs or immunosuppressive agents in the prev.4 weeks
* History of specific immunotherapy with mites
* UV radiation
* Group 4 topical corticosteroids (European classification)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in SCORAD and topical medication consumption | 1 year
  Sccore of atopic dermatitis (SCORAD)

SECONDARY OUTCOMES:
Changes from baseline in SCORAD intensity score, EASI score and change in topical medication consumption | 1 year
  Eczema Area Severity Index (EASI)

OTHER OUTCOMES:
SCORAD extent criteria, index, subjective symptoms, IGA score, oral rescue medication, exacerbation of atopic dermatitis, DLQI, treatment expectation questionnaire | 1 year
  Investigator´s Global Assessment (IGA), Dermatology Life Quality Index (DLQI)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Wolf, PhD, Study Director — ALK-SCHERAX Arzneimittel GmbH; Alexander Kapp, MD, Prof., Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Klinik für Dermatologie und Venerologie, Hanover, Germany